CLINICAL TRIAL: NCT07218458
Title: Enhancing Resilience And Mental Well-Being Through Breathing Practice For Clinical Care Professionals (Breathing Study-Burnout)
Brief Title: A Study Of Resilience And Mental Well-Being Through Breathing Practice For Clinical Care Professionals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Pravesh Sharma, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-009320
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Burnout, Healthcare Workers; Breathing Exercises
Keywords: burnout; breathing
MeSH Terms: conditions — Burnout, Psychological; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breathing Intervention (Experimental): Engaging in self-guided breathing sessions to improve brain circulation and mental well-being.
  Interventions: Behavioral: Structured Breathing

INTERVENTIONS:
Behavioral: Structured Breathing — 15, 30, or 36 minute structured breathing sessions based on personal skill level.

SUMMARY:
The purpose of this study is to assess the immediate and long-term effects of structured breathing on clinical symptoms related to mental health including anxiety, depression, perceived stress, and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthcare professionals at the above-mentioned 4 MCHS sites (Eau Claire, La Crosse, Mankato, Albert Lea).
* Must score ≥40 on Copenhagen Burnout Inventory Q1-6.
* Participants must be physically fit enough to perform light exercise.
* Participants should read and understand English well enough to consent, complete measures, and follow instructions.
* Participants must have access to a smartphone or tablet.

Exclusion Criteria:

* Active primary psychotic disorder or substance use disorder (except nicotine dependence) within the past year.
* Severe or unstable medical condition that could interfere with participation or data collection.
* Active neurological condition (including seizure disorder, traumatic brain injury, or stroke) that could affect cognitive functioning or brain imaging results.
* Chronic lung disease (e.g., COPD, cystic fibrosis) or aneurysm.
* Current pregnancy or planning to become pregnant during the study period

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Assess feasibility of the structured breathing-based intervention among healthcare professionals via ease of recruitment | Enrollment to end of study participation at 4 months.
  This outcome measure will assess whether the structured breathing-based intervention is feasible among healthcare professionals via ease of recruitment reported by study staff.
Assess feasibility of the structured breathing-based intervention among healthcare professionals via retention statistics | Enrollment to end of study participation at 4 months
  This outcome measure will assess the feasibility of the structured breathing-based intervention among healthcare professionals by examining retention rates throughout study duration.
Assess feasibility of the structured breathing-based intervention among healthcare professionals via mobile app engagement metrics | Enrollment to end of study participation at 4 months
  This outcome measure will assess whether the structured breathing-based intervention is feasible among healthcare professionals by analyzing app usage metrics from participants.
Assess feasibility of structured breathing-based intervention among healthcare professionals via Feasibility of Intervention Measure | Enrollment to end of study participation at 4 months
  To assess the feasibility of a structured breathing intervention among healthcare professionals using Feasibility of Intervention Measure (FIM).
  Feasibility of Intervention Measure is a four-item measure of implementation feasibility with scores ranging from 1-5, with higher scores indicating greater feasibility.
Assess appropriateness of structured breathing-based intervention among healthcare professionals | Enrollment to end of study participation at 4 months
  To assess the appropriateness of a structured breathing intervention among healthcare professionals using Intervention Appropriateness Measure (IAM).
  Intervention Appropriateness Measure is a four-item measure with a scale of responses from 1-5, with higher scores indicating greater appropriateness.
Assess acceptability of structured breathing-based intervention among healthcare professionals | From enrollment to the end of study participation at 4 months
  To assess the acceptability of a structured breathing intervention among healthcare professionals utilizing the Acceptability of Intervention Measure (AIM).
  Acceptability of Intervention Measure is a four-item measure with responses from 1-5, with higher scores equating to greater acceptability.
Assess participant satisfaction related to breathing-based intervention | Enrollment to end of study participation at 4 months.
  Participant satisfaction will be assessed through a mixed-methods approach combining quantitative surveys (exit survey) and qualitative participant interviews (4 month in-person visit/interview).

SECONDARY OUTCOMES:
Evaluate intervention adherence, usability, and engagement metrics via mobile application | Enrollment to end of treatment at 4 months.
  To evaluate the breathing intervention adherence, usability, and engagement metrics collected through the mobile application platform. These data will be used to identify barriers and facilitators to digital engagement, assess usability, and inform refinements to the intervention's delivery and technological infrastructure for future large-scale trials.

OTHER OUTCOMES:
Assess the physiological effects of the breathing-based intervention | Enrollment to end of intervention at 4 months. Additional assessments during data analysis period.
  As an exploratory objective, the study will assess the physiological effects of the breathing-based intervention on cerebral oxygenation and local tissue hemodynamics, utilizing functional near-infrared spectroscopy (fNIRS) data performed pre-and-post intervention.
Assess the psychological effects of the breathing-based intervention | Enrollment to end of intervention at 4 months. Additional assessments during data analysis period
  The psychological effects and outcomes will be assessed, using questionnaires completed at specific timepoints throughout the study.
  Questionnaires to include General Health Questionnaire (GHQ), Copenhagen Burnout Inventory (CBI), Generalized Anxiety Disorder scale (GAD), Perceived Stress Scale (PSS), Brief Resilience Scale (BRS).
Assess feasibility of collecting physiological and psychological data | Enrollment to end of study participation at 4 months.
  This exploratory analysis is intended to assess the feasibility of collecting physiological and psychological data from participants, as reported by study staff who are assigned to collect this data.
Assess gathered data to apply to future research | Data analysis period after data collection is complete
  This exploratory analysis will examine study data to identify preliminary trends that can inform the design and power calculations of future definitive trials.

CONTACTS AND LOCATIONS:
Overall Officials: Pravesh Sharma, MD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic Health System-Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health System-Mankato, Mankato, Minnesota
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System-La Crosse, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials